CLINICAL TRIAL: NCT00290433
Title: A Phase II Study of the Efficacy of the HCVIDDOXIL Regimen in Patients With Newly Diagnosed Peripheral T Cell Lymphoma
Brief Title: Efficacy of the HCVIDDOXIL Regimen in Patients With Newly Diagnosed Peripheral T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0004; NCI-2010-00445 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Lymphoma
Keywords: Lymphoma; Peripheral T Cell; HCVIDDOXIL Regimen; ARA-C; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride; Pegylated Liposomal Doxorubicin; Doxorubicin hydrochloride; Doxil; Cyclophosphamide; Cytoxan; Neosar; Dexamethasone; Decadron; Mesna; Methotrexate; Vincristine; G-CSF; Filgrastim; Neupogen
MeSH Terms: conditions — Lymphoma | interventions — Cyclophosphamide; Mesna; Vincristine; Methotrexate; Cytarabine; Dexamethasone; Calcium Dobesilate; Granulocyte Colony-Stimulating Factor; Filgrastim; liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HCVIDDOXIL Regimen (Experimental): Cycle 1: Cyclophosphamide by vein two times a day on Days 1,2, and 3. Mesna by vein nonstop over Days 1 through 3. Pegylated liposomal doxorubicin by vein over 1 hour on Day 2. Vincristine by vein on Days 4 and 11. Dexamethasone by mouth on Days 1 through 4 and 11 through 14.
  Cycle 2: Methotrexate by vein over 2 hours on Day 1 and over 22 hours on day 1. Cytarabine by vein twice a day on Days 2 and 3.
  Interventions: Drug: Cyclophosphamide; Drug: Mesna; Drug: Vincristine; Drug: Methotrexate; Drug: Ara-C; Drug: Dexamethasone; Drug: G-CSF; Drug: Doxil

INTERVENTIONS:
Drug: Cyclophosphamide — Cycle 1: 300 mg/m^2 by vein Over 3 Hours Twice Daily on Days 1, 2, and 3.
  Other Names: Cytoxan; Neosar
Drug: Mesna — Cycle 1: 600 mg/m^2 by vein Continuous Infusion Over Days 1, 2, and 3.
Drug: Vincristine — Cycle 1: 1.4 mg/m^2 by vein On Day 4 and 11.
Drug: Methotrexate — Cycle 1 and 2: 200 mg/m^2 by vein Over 2 Hours on Day 1, followed by 800 mg/m^2 IV Over 22 Hours on Day 1.
Drug: Ara-C — Cycle 1 and 2: 3 Gm/m^2 Over 2 Hours Twice Daily On Days 2 and 3.
  Other Names: Cytarabine; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride
Drug: Dexamethasone — Cycle 1: 40 mg by vein or by mouth daily on Days 1-4 and 11-14.
  Other Names: Decadron
Drug: G-CSF — Cycle 1 and 2: 300 or 480 mcg subcutaneously 24 hours after end of Day 4 vincristine.
  Other Names: Filgrastim; Neupogen
Drug: Doxil — Cycle 1: 25 mg/m^2 by vein Over 1 Hour on Day 2.
  Other Names: Pegylated Liposomal Doxorubicin; Doxorubicin hydrochloride (lipsomal)

SUMMARY:
The goal of this clinical research study is to learn if treatment with two types of chemotherapy combinations can help to control peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
All of the drugs used in this study are commonly used in the treatment of cancer. However, using these drugs in combination is investigational.

During treatment, you will be given two different cycles of chemotherapy, which will be alternated every 21 days.

For Cycle 1, cyclophosphamide will be given by vein two times a day on Days 1,2, and 3. Each dose will take around 3 hours to give. Mesna will be given by vein nonstop over Days 1 through 3. Pegylated liposomal doxorubicin will be given by vein over 1 hour on Day 2. Vincristine will be given by vein on Days 4 and 11. Dexamethasone will be given by mouth on Days 1 through 4 and 11 through 14. Other drugs will be given before, during, and after chemotherapy to help decrease the risk of developing side effects. These drugs may be given by mouth or by injection.

For Cycle 2, methotrexate will be given by vein over 2 hours on Day 1 and over 22 hours on day 1. Cytarabine will be given by vein twice a day on Days 2 and 3. Each dose will take about 2 hours to give. Other drugs will be given before, during, and after treatment to help decrease the risk of developing side effects. These drugs may be given by mouth or by injection.

To help increase the blood counts and help decrease the risk of developing infections, your doctor may decide that treatment with filgrastim is necessary. Filgrastim may be given as once-a-day injections under the skin starting 24 hours after the end of Day 4 vincristine (Cycle 1) and starting 24 hours after the end of Cytarabine (Cycle 2). Your blood counts will be monitored and filgrastim is stopped when the levels become normal.

Cycles 1 and 2 will be alternated every 21 days. Both Cycles 1 and 2 can be given on an outpatient basis if your physician authorizes it. However, if your serum creatinine (blood test) reaches a certain level, Cycle 2 should be given on an inpatient basis.

Depending on how the disease responds, treatment may be stopped after 2,4, or 6 cycles. However, treatment may continue for up to 8 cycles.

During treatment, you will have around 2-3 tablespoons of blood collected at least once a week for routine tests.

After every 2 cycles, tumors will be measured using x-rays or other scans (CT, MRI, etc.) and bone marrow samples will be taken. Heart scans or heart function tests may also be needed if you doctor feels it is necessary.

If the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

After the last cycle of chemotherapy, you will have follow-up exams scheduled. During these exams, you will have a chest x-ray and CT scans of the chest, abdomen (stomach) and pelvis (waist area), and PET scan. You will have blood collected (2-3 tablespoons) for routine tests. If your doctor feels it is necessary, you may also have a sample of bone marrow collected. You may choose to have long-term follow-up exams at M. D. Anderson or with your local physician.

This is an investigational study. All of the study drugs are approved by the FDA for cancer treatment and are commercially available. However, the use of the drugs in combination is experimental. Up to 55 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of previously untreated T-cell Non Hodgkin's Lymphomas and NK lymphomas, with the exception of cluster of differentiation antigen 30 (CD30+) alk1+ T-anaplastic large cell lymphoma (ALCL). Patients with skin involvement alone are also excluded. For patients with skin involvement as part of systemic disease, prior topical treatment only is allowed.
2. Patients with a performance status of 3 or less (Zubrod Scale - see Appendix D).
3. Serum bilirubin </= 1.5 mg/dl and serum creatinine </= 2.0 mg/dl unless due to lymphoma; Absolute neutrophil count (ANC) >/= 1000 mm^3 and platelets >/= 100,000 mm^3 unless due to lymphoma.
4. Cardiac ejection fraction 50% or greater by multigated radionuclide angiography (MUGA) or echocardiogram.
5. Ages 18 and older.
6. Patients must be willing to receive transfusions of blood products.

Exclusion Criteria:

1. Patients with CD30+ alk1+ T-anaplastic large cell lymphoma (ALCL) or patients with skin involvement alone.
2. Pregnancy
3. HIV positive serology
4. Central nervous system (CNS) involvement
5. Co-morbid medical, such as Child's Class C liver cirrhosis, end-stage renal disease, and symptomatic congestive heart failure, or psychiatric illnesses that preclude treatment with intense dose chemotherapy as determined by the primary investigator
6. Concurrent or previous malignancy whose prognosis is poor (<90% probability of survival at 5 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2003-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiro Oki, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Chihara D, Pro B, Loghavi S, Miranda RN, Medeiros LJ, Fanale MA, Hagemeister FB, Fayad LE, Romaguera JE, Samaniego F, Neelapu SS, Younes A, Fowler NH, Rodriguez MA, Wang M, Kwak LW, McLaughlin P, Dang NH, Oki Y. Phase II study of HCVIDD/MA in patients with newly diagnosed peripheral T-cell lymphoma. Br J Haematol. 2015 Nov;171(4):509-16. doi: 10.1111/bjh.13628. Epub 2015 Aug 10. PMID 26260306
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: September 17, 2003 to May 8, 2009. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the 55 participants registered, two participants were found not to be eligible prior to start of study therefore are excluded from trial details.
Groups:
- HCVIDDOXIL Regimen: Cycle 1: Cyclophosphamide 300 mg/m^2 intravenous (IV) twice a day on Days 1-3. Mesna 600 mg/m^2 continuous IV Days 1-3. Doxil 25 mg/m^2 IV over 1 hour on Day 2. Vincristine 1.4 mg/m^2 IV on Days 4 and 11. Dexamethasone 40 mg Iv or oral on Days 1 - 4 and 11 - 14.
  Cycle 2: Methotrexate 200 mg/m^2 over 2 hours on Day 1 and 800 mg/m^2 over 22 hours on day 1. Cytarabine 3 Gm/m^2 IV twice a day on Days 2 and 3.
Period: Overall Study
Arm/Group | HCVIDDOXIL Regimen
Started | 53
Completed | 17
Not Completed | 36
Not completed — Disease Progression | 13
Not completed — Adverse Event | 14
Not completed — Withdrawal by Subject | 1
Not completed — Non-Compliance | 1
Not completed — Congestive Heart Failure | 1
Not completed — Transplant in CR | 5
Not completed — Unrelated Infection/Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | HCVIDDOXIL Regimen
Number analyzed (Participants) | 53
Age, Continuous [Median (Full Range); unit: years] | 54 [20 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: 3 Year Progression-Free Survival Rate
Description: Percentage of participants out of total treated alive with disease progression 3 years following registration. Progression-free survival (PFS) was measured from the date of study registration to the date of documented disease progression or death of any cause.
Time Frame: From registration to disease progression or death, up to 3 years
Population: Of the 53 participants, *6 participants* were not evaluable for response due to either no measurable disease (1) or early departure from study for adverse events (5)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCVIDDOXIL Regimen
Number analyzed (Participants) | 47
percentage of participants | 30 [18 to 44]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the initiation of the regimen through the end of the chemotherapy cycle, up to 3 years.
Arm/Group | HCVIDDOXIL Regimen
Serious Adverse Events (participants affected / at risk) | 1/53
Other Adverse Events (participants affected / at risk) | 46/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCVIDDOXIL Regimen (N=53)
massive cytomegalovirus infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCVIDDOXIL Regimen (N=53)
Neutropenia (Blood and lymphatic system disorders) | 42 (42)
Anemia (Blood and lymphatic system disorders) | 46 (46)
Thrombocytopenia (Blood and lymphatic system disorders) | 46 (46)
Febrile Neutropenia (Blood and lymphatic system disorders) | 21 (21)
Fever (General disorders) | 35 (35)
Infectious Disease (Infections and infestations) | 19 (19)
Fatigue (General disorders) | 40 (40)
Liver Toxicities (Hepatobiliary disorders) | 21 (21)
Constipation (Gastrointestinal disorders) | 19 (19)
Dizziness (Nervous system disorders) | 19 (19)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 (19)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (11)
Mucositis (Respiratory, thoracic and mediastinal disorders) | 16 (16)
Edema (General disorders) | 36 (36)
Rash (Skin and subcutaneous tissue disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes